CLINICAL TRIAL: NCT03378453
Title: Narcolepsy Protect Against Alzheimer's Disease? Protective Role of Low Rates of Orexin on the Occurrence of Intracerebral Amyloid Deposits Characteristic of the Alzheimer's Disease: A Pilot Study
Brief Title: Narcolepsy Protect Against Alzheimer's Disease?
Acronym: PROTECMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9636
Record Dates: First submitted 2016-08-02; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Narcolepsy; Amyloid Pathology
Keywords: Narcolepsy; Alzheimer; Orexin; Amyloid; PET-amyloid imaging
MeSH Terms: conditions — Narcolepsy; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NarCo (Other): Narcolepsy type 1 over 65 years old
  Interventions: Device: PET-scan18F-AV-45
- CoS (Other): Cognitevement healthy controls
  Interventions: Device: PET-scan18F-AV-45

INTERVENTIONS:
Device: PET-scan18F-AV-45 — The PET-scan18F-AV-45 is a PET-scan dedicated to analyze the amyloid load in the brain with the AV45 tracer by the measurement of the mean cortical SuVr
  Arms: NarCo
Device: PET-scan18F-AV-45 — PET-scan18F-AV-45 already done in another protocol MEMENTO-AMYging
  Arms: CoS

SUMMARY:
Links between orexin and amyloid processes have been underlined recently. During the Alzheimer's process an upregulation of the orexin mechanism has been observed. The pathophysiological mechanism of narcolepsy type 1 is linked to orexin deficiency. Thus, the investigators hypothesized that patients with narcolepsy may be protected from amyloid brain lesions, hallmarks of the Alzheimer's process. To test this hypothesis, the investigators analyzed the brain amyloid load measured by PET-scan amyloid brain imaging in patients with narcolepsy type 1 compared to controls without cognitive deficits.

DETAILED DESCRIPTION:
The lack of innovative treatments in Alzheimer' disease (AD) is due to the non-understanding of the pathological process. The investigators need to include the latest concept of the sleep-wake/circadian kinetics of proteins in the brain, the new theory of the wash-out of pathological proteins via the brain glymphatic system during sleep and act at an early stage. New pathways are opened to better understand proteinopathies' processes and to propose new therapeutics interventions. The variations of the production/clearance curves of amyloid in the cerebrospinal fluid (CSF) during circadian rhythms and sleep-wake cycles have been demonstrated in in vivo metabolism experimentations. Suprachiasmatic nucleus damages due to AD may induce circadian regulation dysfunction and secondary sleep/wake cycle alterations. Key sleep/wake cycle neuromediators (Orexin-A, melatonin) are involved in the regulation of brain amyloid levels. The influence of orexin-A signaling on Aβ metabolism in animals and humans was recently highlighted. In rats, orexin-A release shows a 24-h fluctuation similar to that of brain interstitial fluid Aβ. In transgenic mice that overexpress amyloid precursor protein (APP), brain interstitial fluid Aβ concentration increases during wakefulness and after orexin-A infusion. Conversely, it decreases during sleep and after infusion of an orexin-A receptor antagonist6. In transgenic mice that overexpress APP/presenilin1 (PS1), in which the orexin gene is knocked out, a reduction of Aβ pathology was found, possibly caused by changes in sleep time. Orexin-A is linked to Aβ42 in AD and an increase of CSF orexin-A is observed in AD vs. controls, possibly related to sleep deterioration and neurodegeneration.

The narcolepy with cataplexy type 1 is the only disease with a specific orexin deficiency. Montpellier team have previously underlined in 15 patients with narcolepsy type 1 a normal level of Aβ42 in the CSF. The clinical expertise of the narcolepsy center suggested that the frequency of AD in old narcoleptic patients is low. The hypothesis was that patients with narcolepsy type 1 may be protected from amyloid brain lesions, hallmarks of the Alzheimer's process. The objective was to determine whether the brain amyloid load by PET-scan18 F-AV-45 measured with a semi-quantitative analysis (mean cortical SuVr) is lower in patients with narcolepsy type 1 older than 65 years-old than in cognitively normal age- and gender-matched controls.

ELIGIBILITY:
Inclusion criteria:

Narcolepsy group:

* Patients with narcolepsy type 1 older than 65 y.o. with orexin deficiency as required by international diagnosis criteria (ICSD3) with a follow-up in the national reference center for narcolepsy;
* Treated or not with psychostimulant drugs in relation to disease symptoms;
* Patients with CSF samples available or with scheduled lumbar puncture for diagnosis purpose;
* No contra-indications of the PET-scan18F-AV-45
* With a free and informed consent to participate to the study.

Control group:

* Subjects already included in the MEMENTO-AMYging and/or MAPT-AV45 ancillary studies in the memory center with normal cognitive tests after neuropsychological assessments especially in the episodic memory tests and the brain amyloid PET-scan18F-AV-45 data with SuVr measurements.

Exclusion criteria:

* Controls subjects or patients without free and informed consent to participate to the study
* No PET-scan18F-AV-45 data available
* No CSF samples
* Pathologies being life-threatening in a short term
* Patients deprived of freedom by court or administrative order
* Patients living in institution
* Major protected by the Law.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Mean of cortical SuVr based of the PET-scan18F-AV-45 imaging | Upon study completion, an average of one year
  Mean of cortical SuVr based of the PET-scan18F-AV-45 imaging

SECONDARY OUTCOMES:
Mean regional SuVr with PET-scan AV45 | Upon study completion, an average of one year
CSF Amyloid Aβ42 | Upon study completion, an average of one year
  pg/ml
CSF Amyloid Aβ40 | Upon study completion, an average of one year
  pg/ml
CSF Tau protein | Upon study completion, an average of one year
  pg/ml
CSF Orexin concentration | Upon study completion, an average of one year
  pg/ml
Night-time sleep duration | Upon study completion, an average of one year
  Hours/night
Day-time sleep duration | Upon study completion, an average of one year
  Hours/day
Cataplexy | Upon study completion, an average of one year
  Numbers/week
Epworth sleepiness scale (ESS) | Upon study completion, an average of one year
  Score as a number
Beck Depression Inventory (BDI) | Upon study completion, an average of one year
  Score as a number
European Quality of Life Dimension (EQL-5) | Upon study completion, an average of one year
  Score as a number

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Gabelle, MD, PhD, Study Chair — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bateman RJ, Munsell LY, Morris JC, Swarm R, Yarasheski KE, Holtzman DM. Human amyloid-beta synthesis and clearance rates as measured in cerebrospinal fluid in vivo. Nat Med. 2006 Jul;12(7):856-61. doi: 10.1038/nm1438. Epub 2006 Jun 25. PMID 16799555
- [Background] Bateman RJ, Wen G, Morris JC, Holtzman DM. Fluctuations of CSF amyloid-beta levels: implications for a diagnostic and therapeutic biomarker. Neurology. 2007 Feb 27;68(9):666-9. doi: 10.1212/01.wnl.0000256043.50901.e3. PMID 17325273
- [Background] Mawuenyega KG, Sigurdson W, Ovod V, Munsell L, Kasten T, Morris JC, Yarasheski KE, Bateman RJ. Decreased clearance of CNS beta-amyloid in Alzheimer's disease. Science. 2010 Dec 24;330(6012):1774. doi: 10.1126/science.1197623. Epub 2010 Dec 9. PMID 21148344
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Mendelsohn AR, Larrick JW. Sleep facilitates clearance of metabolites from the brain: glymphatic function in aging and neurodegenerative diseases. Rejuvenation Res. 2013 Dec;16(6):518-23. doi: 10.1089/rej.2013.1530. PMID 24199995
- [Background] Kang JE, Lim MM, Bateman RJ, Lee JJ, Smyth LP, Cirrito JR, Fujiki N, Nishino S, Holtzman DM. Amyloid-beta dynamics are regulated by orexin and the sleep-wake cycle. Science. 2009 Nov 13;326(5955):1005-7. doi: 10.1126/science.1180962. Epub 2009 Sep 24. PMID 19779148
- [Background] Coogan AN, Schutova B, Husung S, Furczyk K, Baune BT, Kropp P, Hassler F, Thome J. The circadian system in Alzheimer's disease: disturbances, mechanisms, and opportunities. Biol Psychiatry. 2013 Sep 1;74(5):333-9. doi: 10.1016/j.biopsych.2012.11.021. Epub 2012 Dec 28. PMID 23273723
- [Background] Wu YH, Zhou JN, Van Heerikhuize J, Jockers R, Swaab DF. Decreased MT1 melatonin receptor expression in the suprachiasmatic nucleus in aging and Alzheimer's disease. Neurobiol Aging. 2007 Aug;28(8):1239-47. doi: 10.1016/j.neurobiolaging.2006.06.002. Epub 2006 Jul 11. PMID 16837102
- [Background] Mirmiran M, Swaab DF, Kok JH, Hofman MA, Witting W, Van Gool WA. Circadian rhythms and the suprachiasmatic nucleus in perinatal development, aging and Alzheimer's disease. Prog Brain Res. 1992;93:151-62; discussion 162-3. doi: 10.1016/s0079-6123(08)64570-7. PMID 1480747
- [Background] Hoogendijk WJ, van Someren EJ, Mirmiran M, Hofman MA, Lucassen PJ, Zhou JN, Swaab DF. Circadian rhythm-related behavioral disturbances and structural hypothalamic changes in Alzheimer's disease. Int Psychogeriatr. 1996;8 Suppl 3:245-52; discussion 269-72. doi: 10.1017/s1041610297003426. No abstract available. PMID 9154571
- [Background] Dauvilliers YA, Lehmann S, Jaussent I, Gabelle A. Hypocretin and brain beta-amyloid peptide interactions in cognitive disorders and narcolepsy. Front Aging Neurosci. 2014 Jun 11;6:119. doi: 10.3389/fnagi.2014.00119. eCollection 2014. PMID 24966833
- [Background] Liguori C, Romigi A, Nuccetelli M, Zannino S, Sancesario G, Martorana A, Albanese M, Mercuri NB, Izzi F, Bernardini S, Nitti A, Sancesario GM, Sica F, Marciani MG, Placidi F. Orexinergic system dysregulation, sleep impairment, and cognitive decline in Alzheimer disease. JAMA Neurol. 2014 Dec;71(12):1498-505. doi: 10.1001/jamaneurol.2014.2510. PMID 25322206
- [Background] Slats D, Claassen JA, Verbeek MM, Overeem S. Reciprocal interactions between sleep, circadian rhythms and Alzheimer's disease: focus on the role of hypocretin and melatonin. Ageing Res Rev. 2013 Jan;12(1):188-200. doi: 10.1016/j.arr.2012.04.003. Epub 2012 Apr 30. PMID 22575905
- [Background] Yoshida Y, Fujiki N, Nakajima T, Ripley B, Matsumura H, Yoneda H, Mignot E, Nishino S. Fluctuation of extracellular hypocretin-1 (orexin A) levels in the rat in relation to the light-dark cycle and sleep-wake activities. Eur J Neurosci. 2001 Oct;14(7):1075-81. doi: 10.1046/j.0953-816x.2001.01725.x. PMID 11683899
- [Background] Roh JH, Jiang H, Finn MB, Stewart FR, Mahan TE, Cirrito JR, Heda A, Snider BJ, Li M, Yanagisawa M, de Lecea L, Holtzman DM. Potential role of orexin and sleep modulation in the pathogenesis of Alzheimer's disease. J Exp Med. 2014 Dec 15;211(13):2487-96. doi: 10.1084/jem.20141788. Epub 2014 Nov 24. PMID 25422493
- [Background] Wennstrom M, Londos E, Minthon L, Nielsen HM. Altered CSF orexin and alpha-synuclein levels in dementia patients. J Alzheimers Dis. 2012;29(1):125-32. doi: 10.3233/JAD-2012-111655. PMID 22207004
- [Derived] Gabelle A, Jaussent I, Bouallegue FB, Lehmann S, Lopez R, Barateau L, Grasselli C, Pesenti C, de Verbizier D, Beziat S, Mariano-Goulart D, Carlander B, Dauvilliers Y; Alzheimer's Disease Neuroimaging Initiative; Multi-Domain Intervention Alzheimer's Prevention Trial study groups. Reduced brain amyloid burden in elderly patients with narcolepsy type 1. Ann Neurol. 2019 Jan;85(1):74-83. doi: 10.1002/ana.25373. Epub 2018 Dec 19. PMID 30387527